CLINICAL TRIAL: NCT00333853
Title: Self-Monitoring of Blood Glucose Study#1: The Ability of People With Diabetes to Use OneTouch(R) Ultrasmart(tm) to Improve Glycemic Control Through Behavioral and Therapeutic Changes
Brief Title: Self-Monitoring of Blood Glucose Study#1: The Ability of People With Diabetes to Use OneTouch(R) Ultrasmart(tm)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: LifeScan (Industry)
Responsible Party: LifeScan, Inc.
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: DDI 70-97017-17
Record Dates: First submitted 2006-06-02; First posted 2006-06-06 (Estimated); Last update posted 2008-05-13 (Estimated); Status verified 2008-05

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: OneTouch(r) UltraSmart(r)

SUMMARY:
Insulin therapy requires monitoring and frequent review of glucose levels to optimize dosing. Effective presentation and data analysis are essential. We examined HbA1c changes using the OneTouch(R) UltraSmart(R) System (Test Group), an integrated glucose meter and electronic logbook, compared to established meters with paper logbooks (Control Group).

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects with type 1 or type 2 insulin-treated diabetes mellitus with a baseline HbA1c greater than or equal to 8.0%.
* The lower age limit for pediatric subjects was at the discretion of the pediatric investigators and their Institutional Review Board (IRBs).
* The upper age limit for pediatric subjects was 20 years (i.e., not having reached their 21st birthday on date of enrollment).
* Subjects must have monitored blood glucose at least 2 times per day. - Subject's current blood glucose meter has download capability, however, the subject did not routinely use this capability on his/her own.

Exclusion Criteria:

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 250
Dates: Start 2003-08; Study Completion 2005-06

PRIMARY OUTCOMES:
Hemoglobin A1c (HbA1c)

SECONDARY OUTCOMES:
Measured hypoglycemia

CONTACTS AND LOCATIONS:
Overall Officials: Lori Laffel, MD, MPH, Principal Investigator — Joslin Diabetes Center
Locations (7):
- United States (7):
  - Diabetes and Endocrine Associates, La Jolla, California
  - Children's Hospital, Los Angeles, Los Angeles, California
  - University of Miami Miller School of Medicine, Miami, Florida
  - University of Maryland School of Medicine, Baltimore, Maryland
  - Joslin Diabetes Center, Boston, Massachusetts
  - Washington University School of Medicine, St Louis, Missouri
  - Radiant Research, Portland, Oregon

REFERENCES:
- [Result] Laffel LM, Hsu WC, McGill JB, Meneghini L, Volkening LK. Continued use of an integrated meter with electronic logbook maintains improvements in glycemic control beyond a randomized, controlled trial. Diabetes Technol Ther. 2007 Jun;9(3):254-64. doi: 10.1089/dia.2006.0021. PMID 17561796